CLINICAL TRIAL: NCT03215953
Title: Offloading Interventions for Diabetic Foot Problems in Upper Egypt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammad Hasan AbdEllah, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OIDFUE001
Record Dates: First submitted 2017-07-09; First posted 2017-07-12 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: offloading; plantar pressure; Diabetic Foot Ulcer; removable offloading device; adherence
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): cast shoe plus standard wound care
  Interventions: Device: cast shoe
- Group B (Active Comparator): removable walker plus standard wound care
  Interventions: Device: removable walker

INTERVENTIONS:
Device: cast shoe — ankle-high, custom-made, well-moulded cast shoe
  Arms: Group A
Device: removable walker — Prefabricated especially designed for relieving load on the foot
  Arms: Group B

SUMMARY:
Offloading is the concept of relieving pressure to help prevent/cure plantar ulcers, especially in diabetic patients. Many forms of offloading are available, with many limitations to apply in clinical practice. In this study, the investigators compare cast shoe with removable walker considering effectiveness, complications, compliance and patient's appreciation.

DETAILED DESCRIPTION:
Abnormal glucose metabolism gradually impairs sensation in both feet. Impaired sensation leads to recurrent attacks of inflammation "acute Charcot arthritis". Eventually, the foot becomes deformed with abnormal shape of the plantar surface. During walking, both neuropathy and deformities cause abnormal distribution of pressure with some points in the plantar surface having a very high pressure. This high pressure leads to skin ulceration "pressure ulcer". These pressure ulcers tend to be recurrent or chronic as long as the problem of high pressure is not resolved.

Offloading techniques are pressure-relieving interventions that redistribute body weight over the plantar surface. Areas with high pressure which are at high risk of ulceration, are treated to decrease pressure and cure ulcers.

The diabetic foot clinic at Assiut university hospital provides patients with necessary care to avoid the single most fearsome enemy, amputation. This clinic currently provides many offloading options based on expert opinion, and there is an urgent need to have a well-balanced view supported by evidence, considering both the physician and the patient.

The investigators' project is to conduct a series of trials to guide policies concerned with diabetic foot problems, OIDFUA. This study will compare cast shoe with removable walker, as different offloading options to cure diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes, loss of protective sensation, forefoot pressure ulcer

Exclusion Criteria:

* Ankle/Brachial index less than 0.7, severe infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of mean ulcer radius | 6 months
  Mean ulcer radius is √(area/π)
Non-severe adverse events related to use of offloading device | 6 months
  abrasions, maceration, fungal infection, or falls that the patient relates to device use Non-severe means resolved within two weeks and device use resumed
Severe adverse events related to use of offloading device | 6 months
  new ulcer, acute Charcot episode, foot infection, or amputation that the patient relates to device use

SECONDARY OUTCOMES:
Adherence | 6 months
  patient's subjective estimation of days per week and hours per day wearing the device of the total days/hours
Perception | 6 months
  patient's own opinion regarding his overall appreciation as a visual analogue score
severity of pain | 6 months
  patient's own opinion regarding pain as a visual analogue score
Mobility | 6 months
  patient's own opinion regarding limitation of mobility as visual analogue score
Lifestyle limitation | 6 months
  patient's own opinion regarding how far the device interferes with his daily activities by naming the activities that needed more effort, e.g. bathing, or stopped, e.g. going to work.

CONTACTS AND LOCATIONS:
Overall Officials: Walaa A Khalifa, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bus SA, Armstrong DG, van Deursen RW, Lewis JE, Caravaggi CF, Cavanagh PR; International Working Group on the Diabetic Foot. IWGDF guidance on footwear and offloading interventions to prevent and heal foot ulcers in patients with diabetes. Diabetes Metab Res Rev. 2016 Jan;32 Suppl 1:25-36. doi: 10.1002/dmrr.2697. No abstract available. PMID 26813614